CLINICAL TRIAL: NCT06018909
Title: The Effect of Cognitive-Behavioral Intervention Package on Peripheral Venous Cannulation Pain and Anxiety in Children: A Randomized Controlled Trial
Brief Title: The Effect of Cognitive-Behavioral Intervention Package on Procedural Pain and Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aynur Aytekin Ozdemir (Other)
Responsible Party: Sponsor-Investigator, Aynur Aytekin Ozdemir, Professor, Istanbul Medeniyet University
Organization: Istanbul Medeniyet University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018-3/20
Record Dates: First submitted 2023-08-21; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Procedural Anxiety; Procedural Pain
Keywords: Anxiety; Children; Procedural pain; Cognitive-behavioral interventions
MeSH Terms: conditions — Pain, Procedural; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants were randomized into the experimental and control groups using a block randomization method. The variables of age (7-9 and 10-12 years), gender (girls and boys), and fear of procedure (yes and no) were used for block randomization.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-Behavioral Interventions Package Group (Experimental): Participants received CBIP. CBIP included procedural preparation and information, distraction, suggestions, parent training and positive reinforcement.
  Interventions: Behavioral: Cognitive-Behavioral Interventions Package
- Control (No Intervention): The control group received the routine peripheral venous cannulation procedure.

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Interventions Package — CBIP was developed by researchers in line with the relevant literature according to the developmental characteristics of children. Opinions were obtained from experts in the field of pediatrics or psychiatric nursing regarding CBIP. CBIP consisted of cognitive and behavioral practices to prevent/reduce procedural pain and anxiety.
  Arms: Cognitive-Behavioral Interventions Package Group

SUMMARY:
This study investigated the effect of cognitive-behavioral interventions package (CBIP) on pain and anxiety related to peripheral venous cannulation (PVC) in children aged 7-12 years.

DETAILED DESCRIPTION:
The International Guide to Pediatric Anesthesia (Good Practice in Postoperative and Procedural Pain) recommends pharmacological and nonpharmacological methods to effectively manage and prevent acute procedural pain in children. Nonpharmacological methods alone or in combination with pharmacological methods help reduce pain, and therefore, have become popular especially in recent years. For pain management, nonpharmacological methods are easy to use, and cost- and time-effective methods with no side effects. Studies have evaluated a large number of pharmacological and nonpharmacological interventions for procedural pain management in children. However, most of those interventions are not used by healthcare professionals because they are expensive, time-consuming or hard to use. Therefore, easy-to-use, practical, non-invasive, cost-effective, and reusable nonpharmacological methods can be used especially in acute settings. Cognitive-behavioral interventions, one of the non-pharmacological methods used to minimize pain and anxiety related to painful medical procedures in children are promising.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 7 to 12 years
* be literate
* requiring peripheral venous cannulation procedure

Exclusion Criteria:

* had chronic diseases
* had neuro-developmentally delayed
* had visual, audio, or speech impairments
* were hospital stay for treatment in the past three years
* had a history of sedative, analgesic or narcotic use within 24 hours before procedure

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale: VAS | Through painful procedure completion, an average of 10 minutes
  The VAS is used to measure and monitor pain intensity. VAS is a 10 cm or 100 mm long horizontal or vertical line with anchor statements "no pain or pain at its least" at the left-most end and "unbearable pain or worst pain imaginable" at the right-most end. The participant is asked to mark a point on the line that best represents their pain level. The VAS score is determined by measuring the distance of the mark from the left end of the line. VAS is an easy-to-understand and easy-to-measure scale for children aged 7 and over.
Wong-Baker FACES Pain Rating Scale: WB-FACES | Through painful procedure completion, an average of 10 minutes
  The scale is used to diagnose pain in children aged 3-18 years. It consists of six facial expressions, each one representing an increasing degree of pain scored on a scale 0 to 5 from left to right. The first face is a happy face representing "no pain=0" while the last face is a crying face representing "the worst pain imaginable=5". Higher scores indicate low pain tolerance. Participants are asked to choose the facial expression that best represents their pain.
Children's Fear Scale: CFS | Through painful procedure completion, an average of 10 minutes
  The CFS was developed to measure fear and anxiety in children. It consists of five facial expressions that represent a range from neutral to extreme fear. It is scored between 0 and 4. Both researchers and family members can use the CFS to measure fear and anxiety in children before and during procedures.
State-Trait Anxiety Inventory for Children-State Form (STAIC-State) | Through painful procedure completion, an average of 10 minutes
  STAIC was designed as a research tool for the study of anxiety in 9- to 12-year-old children as well as in younger or older children depending on their reading ability. The widely used STAIC-State Form includes 20-item self-report scale situational variation. In the STAIC-State Form, the children were asked to evaluate how they felt "that moment" and mark one of the relevant choices. When the presence of these feelings is stated as "much" by the child, the highest score is 3; and when it is not stated, the lowest score is 1.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Aytekin Özdemir, PhD, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Result] Hsieh YC, Cheng SF, Tsay PK, Su WJ, Cho YH, Chen CW. Effectiveness of Cognitive-behavioral Program on Pain and Fear in School-aged Children Undergoing Intravenous Placement. Asian Nurs Res (Korean Soc Nurs Sci). 2017 Dec;11(4):261-267. doi: 10.1016/j.anr.2017.10.002. Epub 2017 Oct 26. PMID 29290273
- [Result] McCarthy AM, Cool VA, Hanrahan K. Cognitive behavioral interventions for children during painful procedures: research challenges and program development. J Pediatr Nurs. 1998 Feb;13(1):55-63. doi: 10.1016/S0882-5963(98)80069-9. PMID 9503767
- [Result] Uman LS, Birnie KA, Noel M, Parker JA, Chambers CT, McGrath PJ, Kisely SR. Psychological interventions for needle-related procedural pain and distress in children and adolescents. Cochrane Database Syst Rev. 2013 Oct 10;(10):CD005179. doi: 10.1002/14651858.CD005179.pub3. PMID 24108531
- [Result] Uman LS, Chambers CT, McGrath PJ, Kisely S. A systematic review of randomized controlled trials examining psychological interventions for needle-related procedural pain and distress in children and adolescents: an abbreviated cochrane review. J Pediatr Psychol. 2008 Sep;33(8):842-54. doi: 10.1093/jpepsy/jsn031. Epub 2008 Apr 2. PMID 18387963
- [Result] Yilmaz Kurt F, Aytekin Ozdemir A, Atay S. The Effects of Two Methods on Venipuncture Pain in Children: Procedural Restraint and Cognitive-Behavioral Intervention Package. Pain Manag Nurs. 2020 Dec;21(6):594-600. doi: 10.1016/j.pmn.2019.09.002. Epub 2019 Oct 15. PMID 31628067
- [Derived] Demir Imamoglu Z, Aytekin Ozdemir A. The effect of a cognitive behavioural intervention package on peripheral venous cannulation pain, fear and anxiety in Paediatric patients: A randomised controlled trial. J Pediatr Nurs. 2024 May-Jun;76:192-198. doi: 10.1016/j.pedn.2024.02.003. Epub 2024 Feb 28. PMID 38417207